CLINICAL TRIAL: NCT03743857
Title: Effects of Improvement of the Ankle Joint Range on Balance in the Elderly: Randomized Controlled Trial
Brief Title: Effects of Improvement of the Ankle Joint Range on Balance in the Elderly.
Acronym: ANKLE_ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHG03
Record Dates: First submitted 2018-11-11; First posted 2018-11-16 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Aging Problems
Keywords: Ankle; Balance; Manual Therapy; Older Adult
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Experimental): 6 sessions of ankle manual therapy
  Interventions: Procedure: Manual Therapy
- Control (No Intervention): No intervention

INTERVENTIONS:
Procedure: Manual Therapy — AP ankle mobilization
  Arms: Manual Therapy

SUMMARY:
The effects of aging on the ankle joint will contribute negatively to balance in the elderly. Manual therapy is a technique that is usually used to treat ankle arthrokinematics, although there is little literature on this population. This study seeks to investigate the effects that a mobilization on the ankle will produce in order to improve its joint range and if the balance of the older adult improves after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or more

Exclusion Criteria:

* Do not sign the consent
* No acute pathology (3 months)
* Vestibular pathology
* CNS disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Test Up and Go | Change from baseline to day 21
  It is a test in which the functional mobility of the participant is measured.
One Leg Balance Test | Change from baseline to day 21
  The time that the participant can be with monopodal support is measured
Functional Reach Test | Change from baseline to day 21
  It measures the ability to move the center of gravity forward without losing balance.
Analysis of Center of Pressure | Change from baseline to day 21
  Measurement of the displacement of the center of pressures using a Pressure Platform.

SECONDARY OUTCOMES:
Active ankle range of movement | Change from baseline to day 21
  Measurement of the total active joint range of the ankle in discharge with a goniometer.
Weight Bearing Dorsiflexion Lunge Test | Change from baseline to day 21
  Measurement of dorsiflexion of the ankle under load with an inclinometer.
Falls Efficacy Scale | Change from baseline to day 21
  Scale that measures the worry of suffering a fall.
Assessment of ankle plantar flexion muscle strength | Change from baseline to day 21
  Measurement of the strength of the plantar flexion of the ankle with a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, Principal Investigator — Study Principal Investigator
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided